CLINICAL TRIAL: NCT04763473
Title: AVocAdo Extract to Improve gLycemia in Individuals With Obesity (AVAIL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Adelaide (Other)
Collaborators: Isagenix International LLC (Industry); Commonwealth Scientific and Industrial Research Organisation, Australia (Other Government); Prolongevity Technologies (Industry)
Responsible Party: Principal Investigator, A/Prof Leonie Heilbronn, Associate Professor, University of Adelaide
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H-2020-248
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Obesity
Keywords: Obesity; Avocado extract; Cardiometabolic health
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants will consume 10 grams of corn meal daily for 12 weeks.
  Interventions: Dietary Supplement: Placebo
- Avocado extract (Experimental): Participants will consume 10 grams of freeze dried avocado daily for 12 weeks.
  Interventions: Dietary Supplement: Avocado extract

INTERVENTIONS:
Dietary Supplement: Avocado extract — Participants will consume 10 grams of freeze dried avocado daily for 12 weeks.
  Arms: Avocado extract
Dietary Supplement: Placebo — Participants will consume 10 grams of corn meal daily for 12 weeks.
  Arms: Placebo

SUMMARY:
This two-arm, double blind, randomized clinical trial will compare the effect of an avocado extract, compared to placebo, on cardiometabolic outcomes in adults with obesity.

DETAILED DESCRIPTION:
Sixty eligible participants will be stratified by sex and randomly assigned to placebo or avocado extract supplementation group for 12 weeks. Metabolic testing will be performed at baseline, and at the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 25 - 65 years old
* Waist circumference (>94cm in men and >80cm in women)
* BMI 30 - 40 kg/m2
* Willingness to provide written informed consent and willingness to participate and comply with the study

Exclusion Criteria:

* Women planning pregnancy during the course of the study or 3 months after completion of the study, or who are lactating
* Individuals diagnosed with type 1 or type 2 diabetes mellitus, liver or kidney diseases, neoplastic disease in the previous 3 years, chronic gastrointestinal disorders (including inflammatory bowel disease and celiac), cardiovascular event in the previous 6 months, or any other condition deemed unstable
* Biochemical abnormalities or evidence at screening of disease including elevated liver enzymes ALT and/or AST >3 times normal range limit
* Not weight-stable (< 5 % fluctuation in their body weight for past 6-months at study entry).
* Current or recent (within 12 months) treatment with medication used to lower blood glucose or antidiabetic medications (metformin, sulfonylureas, glucagon-like peptide-1 (GLP-1) analogues [i.e. exenatide], thiazolidinediones or DPP-IV inhibitors [i.e. 'gliptins']), medications affecting weight, appetite or gut motility (i.e. domperidone, cisapride, orlistat, phentermine, topiramate). Participants who are taking stable doses (i.e. > 12 months) of androgenic medications (i.e. testosterone), thyroxine, corticosteroids, anti-depressants (selective serotonin reuptake inhibitors), anti-hypertensives (ace-inhibitors, calcium channel blockers, beta-blockers, diuretics) and lipid lowering medications (statins, fibrates) will not be excluded.
* Participants who have had bariatric surgery
* Participants with conditions that may interfere with the ability to understand the requirements of the study.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-08-11 (Actual)

PRIMARY OUTCOMES:
Glycemic response | 12 weeks
  Change in glucose area under the curve (AUC) in response to 75 g oral glucose tolerance test

SECONDARY OUTCOMES:
Fasting glucose | 12 weeks
  Change in fasting glucose
Fasting insulin | 12 weeks
  Change in fasting insulin
Postprandial insulin | 12 weeks
  Change in insulin AUC in response to 75g oral glucose tolerance test
Homeostatic model assessment of insulin resistance (HOMA-IR) | 12 weeks
  Change in HOMA-IR
Body weight | 12 weeks
  Change in body weight
Waist circumference | 12 weeks
  Change in waist circumference
Body composition | 12 weeks
  Change in body composition assessed by dual-energy X-ray absorptiometry (DEXA)
Blood pressure | 12 weeks
  Change in systolic and diastolic blood pressure
Blood lipids | 12 weeks
  Change in total cholesterol, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol and triglycerides
C-reactive protein | 12 weeks
  Change in blood C-reactive protein
Oxidative stress | 12 weeks
  Change in blood isoprostane
Autophagy | 12 weeks
  Changes in blood mRNA levels of autophagy markers

CONTACTS AND LOCATIONS:
Overall Officials: Leonie Heilbronn, Principal Investigator — The University of Adelaide
Locations (1):
- The University of Adelaide, Adelaide, South Australia, Australia